CLINICAL TRIAL: NCT05297318
Title: Applying Hypotension Prediction Index Guidance for Prevention of Intraoperative Hypotension in Older Patients Undergoing Major Gastrointestinal Surgery: A Randomized Trial
Brief Title: HPI in Older Patients Undergoing Major Gastrointestinal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 202112225DIND
Record Dates: First submitted 2022-03-17; First posted 2022-03-28 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2022-03

CONDITIONS: the Severity and Duration of Intraoperative Hypotension

STUDY DESIGN:
Intervention Model Description: The patients receive elective major gastrointestinal surgery with older than 65 years old. These patients have divided into two groups, including with/without HPI guided. The intraoperative hypotension incidence has been measured.
Who Masked: Participant, Care Provider
Masking Description: patients and care providers did not know the whether the hypotension prediction index use during the operation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hypotension prediction index guided (Experimental): Patients receiving hypotension prediction index guided. In this group, they will be alerted when the index exceeded 85 (range 0 to 100) indicating the later occurrence of MAP< 65mmHg for at least minutes and a treatment protocol based on advanced hemodynamic parameters recommended vasopressor or inotrope, fluid administration, or observation.
  Interventions: Device: hypotension prediction index guided
- without hypotesion prediction index guided (Sham Comparator): Patients will receive usual care during the operation without hypotension prediction index alerted.
  Interventions: Other: without hypotesion prediction index guided

INTERVENTIONS:
Device: hypotension prediction index guided — patients receiving hypotension prediction index monitoring and let the anesthesiologist' alerted the coming intraoperatiobe hypotension
  Arms: hypotension prediction index guided
Other: without hypotesion prediction index guided — patients receiving usual care without hypotension prediction index monitoring but with usual arterial line care
  Arms: without hypotesion prediction index guided

SUMMARY:
The incidence of intraoperative hypotension was 91%. The increasing incidence of intraoperative hypotension would increase the risk of postoperative complications, such as postoperative arrythmia, stroke or acute kidney injury. Major gastrointestinal surgery is a major surgery. Older patients usually have many comorbidity, such as hypertension or cardiovascular disease. Prevention intraoperative hypotension is an important issue. Hypotension prediction index (HPI) could give the clinician pre-alarm of hypotension (mean arterial pressure (MAP)<65mmHg). In this study, we aimed to investigate whether HPI could prevent the intraoperative hypotension happened in patients receive elective major gastrointestinal surgery with older than 65 years old.

DETAILED DESCRIPTION:
Background: the incidence of intraoperative hypotension was 91%. The increasing incidence of intraoperative hypotension would increase the risk of postoperative complications, such as postoperative arrythmia, stroke or acute kidney injury. Major gastrointestinal surgery is a major surgery. Older patients usually have many comorbidity, such as hypertension or cardiovascular disease. Prevention intraoperative hypotension is an important issue. Hypotension prediction index (HPI) could give the clinician pre-alarm of hypotension (mean arterial pressure (MAP)<65mmHg).

Objectives: to investigate whether HPI could prevent the intraoperative hypotension happened.

Patients and methods: The patients receive elective major gastrointestinal surgery with older than 65 years old. These patients have divided into two groups, including with/without HPI guided. The intraoperative hypotension incidence has been measured.

Expected result: The HPI would significantly decrease the intraoperative hypotension incidence.

ELIGIBILITY:
Inclusion Criteria:

* the age of patients>=65 years old
* patients receivedd major gastrointestinal surgery

Exclusion Criteria:

* patients with major organ dysfunction, such as severe arrythmia, heart failure, under hemodialysis

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2023-10-02 (Actual); Study Completion 2023-11-05 (Actual)

PRIMARY OUTCOMES:
Time-weighted average mean arterial pressure less than 65 mmHg | preoperative and postoperative 30 days
  A higher data of time-weighted average mean arterial pressure less than 65 mmHg indicates severe and longer intraoperative hypotension

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Jun Lai, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Chih-Jun Lai, Taipei, Zhongzheng, Taiwan

IPD SHARING:
Plan to Share IPD: No
ethical issue: patients' privacy